CLINICAL TRIAL: NCT03816995
Title: A Novel Wound Retractor Combining Continuous Irrigation and Barrier Protection Reduces Incisional Contamination and Surgical Site Infection in Colorectal Surgery
Brief Title: Prospective, Randomized, Parallel-arm Clinical Trial of CleanCision or Alexis O in Elective Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scott Steele (Other)
Collaborators: Prescient Surgical (Industry)
Responsible Party: Sponsor-Investigator, Scott Steele, President, Main Campus Submarket, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-1346
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Surgery
Keywords: wound irrigation; cleancision; colorectal surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Alexis O Wound Protector (Active Comparator): Participants will undergo standard surgical procedure using the Alexis O wound protector.
  Interventions: Device: Alexis O Wound Protector
- CleanCision Wound Protector (Experimental): Participants will undergo standard surgical procedure using the CleanCision Wound Retraction and Protection System
  Interventions: Device: CleanCision Wound Retraction and Protection System

INTERVENTIONS:
Device: CleanCision Wound Retraction and Protection System — wound retraction and irrigation
  Arms: CleanCision Wound Protector
Device: Alexis O Wound Protector — wound retraction
  Arms: Alexis O Wound Protector

SUMMARY:
Surgical site infection (SSI) remains a problem in colorectal surgery. Strategies to reduce the incidence of SSI following colorectal surgery are important to improve overall patient outcomes, reduce healthcare-associated costs and provide value-based healthcare to surgical patients.

Preventing contamination of the wound through the use of barrier wound protectors or intraoperative wound irrigation has shown significant promise individually and is an ongoing focus to reduce wound infections SSI.

DETAILED DESCRIPTION:
Surgical site infection (SSI) remains a persistent and morbid problem in colorectal surgery with published rates ranging from 7 to 25%. The negative outcomes of SSI are well reported and include a significant increase in morbidity, length of hospital stay, readmissions and healthcare-associated cost. Therefore, strategies to reduce the incidence of SSI following colorectal surgery are important to improve overall patient outcomes, reduce healthcare-associated costs and provide value-based healthcare to surgical patients.

Key to the pathogenesis of SSI is the degree of bacterial contamination of the surgical wound. Preventing contamination of the wound or reducing the bacterial load through the use of barrier wound protectors or intraoperative wound irrigation has shown significant promise individually and is an ongoing strategic focus to reduce wound infections after surgery.

The usage of intraoperative wound irrigation has been shown to significantly reduce the risk of SSI via multiple RTC. A surgical device that combines continuous wound irrigation and barrier protection will have an important SSI prevention advantage.

CleanCision is a recently developed apparatus that serves this purpose and was found to reduce bacterial wound contamination in preclinical and clinical trials.

This study aims to investigate the effect of using CleanCision wound protector on the rates of postoperative Surgical Site Infections in comparison to the current wound protector (Alexis O) being used at our institute.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years old and above.
2. Elective colorectal surgery with a planned resection including open or laparoscopic surgeries.
3. Clean -contaminated, contaminated and dirty wounds per the definition above.
4. Patients undergoing Standard of care SSI reduction bundle including Prophylactic AB and mechanical bowel preparation.
5. Anticipated incision length of 3-17 cm

Exclusion Criteria:

1. Patients younger than 18 years old.
2. Patients with a preexisting stoma.
3. Patients with prior laparotomy within 15 days.
4. Patients with an active infection or systemic antibiotic therapy within 1 week prior to surgery with the exception of preoperative antimicrobial prophylaxis.
5. Emergent/ urgent surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Steele, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walz JM, Paterson CA, Seligowski JM, Heard SO. Surgical site infection following bowel surgery: a retrospective analysis of 1446 patients. Arch Surg. 2006 Oct;141(10):1014-8; discussion 1018. doi: 10.1001/archsurg.141.10.1014. PMID 17043280
- [Background] Smith RL, Bohl JK, McElearney ST, Friel CM, Barclay MM, Sawyer RG, Foley EF. Wound infection after elective colorectal resection. Ann Surg. 2004 May;239(5):599-605; discussion 605-7. doi: 10.1097/01.sla.0000124292.21605.99. PMID 15082963
- [Background] Konishi T, Watanabe T, Kishimoto J, Nagawa H. Elective colon and rectal surgery differ in risk factors for wound infection: results of prospective surveillance. Ann Surg. 2006 Nov;244(5):758-63. doi: 10.1097/01.sla.0000219017.78611.49. PMID 17060769
- [Background] de Oliveira AC, Ciosak SI, Ferraz EM, Grinbaum RS. Surgical site infection in patients submitted to digestive surgery: risk prediction and the NNIS risk index. Am J Infect Control. 2006 May;34(4):201-7. doi: 10.1016/j.ajic.2005.12.011. PMID 16679177
- [Background] Fujii S, Tsukamoto M, Fukushima Y, Shimada R, Okamoto K, Tsuchiya T, Nozawa K, Matsuda K, Hashiguchi Y. Systematic review of laparoscopic vs open surgery for colorectal cancer in elderly patients. World J Gastrointest Oncol. 2016 Jul 15;8(7):573-82. doi: 10.4251/wjgo.v8.i7.573. PMID 27559437
- [Background] Serra-Aracil X, Garcia-Domingo MI, Pares D, Espin-Basany E, Biondo S, Guirao X, Orrego C, Sitges-Serra A. Surgical site infection in elective operations for colorectal cancer after the application of preventive measures. Arch Surg. 2011 May;146(5):606-12. doi: 10.1001/archsurg.2011.90. PMID 21576613
- [Background] de Lissovoy G, Fraeman K, Hutchins V, Murphy D, Song D, Vaughn BB. Surgical site infection: incidence and impact on hospital utilization and treatment costs. Am J Infect Control. 2009 Jun;37(5):387-397. doi: 10.1016/j.ajic.2008.12.010. Epub 2009 Apr 23. PMID 19398246
- [Background] Tanner J, Khan D, Aplin C, Ball J, Thomas M, Bankart J. Post-discharge surveillance to identify colorectal surgical site infection rates and related costs. J Hosp Infect. 2009 Jul;72(3):243-50. doi: 10.1016/j.jhin.2009.03.021. Epub 2009 May 15. PMID 19446918
- [Background] Wick EC, Vogel JD, Church JM, Remzi F, Fazio VW. Surgical site infections in a "high outlier" institution: are colorectal surgeons to blame? Dis Colon Rectum. 2009 Mar;52(3):374-9. doi: 10.1007/DCR.0b013e31819a5e45. PMID 19333034
- [Background] Gorgun E, Rencuzogullari A, Ozben V, Stocchi L, Fraser T, Benlice C, Hull T. An Effective Bundled Approach Reduces Surgical Site Infections in a High-Outlier Colorectal Unit. Dis Colon Rectum. 2018 Jan;61(1):89-98. doi: 10.1097/DCR.0000000000000929. PMID 29215475
- [Background] Sajid MS, Rathore MA, Sains P, Singh KK. A systematic review of clinical effectiveness of wound edge protector devices in reducing surgical site infections in patients undergoing abdominal surgery. Updates Surg. 2017 Mar;69(1):21-28. doi: 10.1007/s13304-017-0415-2. Epub 2017 Jan 25. PMID 28124278
- [Background] Ruiz-Tovar J, Santos J, Arroyo A, Llavero C, Armananzas L, Lopez-Delgado A, Frangi A, Alcaide MJ, Candela F, Calpena R. Effect of peritoneal lavage with clindamycin-gentamicin solution on infections after elective colorectal cancer surgery. J Am Coll Surg. 2012 Feb;214(2):202-7. doi: 10.1016/j.jamcollsurg.2011.10.014. PMID 22265220
- [Background] Mueller TC, Loos M, Haller B, Mihaljevic AL, Nitsche U, Wilhelm D, Friess H, Kleeff J, Bader FG. Intra-operative wound irrigation to reduce surgical site infections after abdominal surgery: a systematic review and meta-analysis. Langenbecks Arch Surg. 2015 Feb;400(2):167-81. doi: 10.1007/s00423-015-1279-x. Epub 2015 Feb 14. PMID 25681239
- [Background] Solomkin J, Gastmeier P, Bischoff P, Latif A, Berenholtz S, Egger M, Allegranzi B. WHO Guidelines to prevent surgical site infections-Authors' reply. Lancet Infect Dis. 2017 Mar;17(3):262-264. doi: 10.1016/S1473-3099(17)30081-6. Epub 2017 Feb 23. No abstract available. PMID 28244389
- [Background] Papaconstantinou HT, Ricciardi R, Margolin DA, Bergamaschi R, Moesinger RC, Lichliter WE, Birnbaum EH. A Novel Wound Retractor Combining Continuous Irrigation and Barrier Protection Reduces Incisional Contamination in Colorectal Surgery. World J Surg. 2018 Sep;42(9):3000-3007. doi: 10.1007/s00268-018-4568-z. PMID 29523908

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alexis O Wound Protector | CleanCision Wound Protector
Started | 351 | 351
Completed | 327 | 318
Not Completed | 24 | 33
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Cancelled Surgery | 8 | 12
Not completed — No wound protector used | 11 | 17
Not completed — Protocol Violation | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alexis O Wound Protector | CleanCision Wound Protector | Total
Number analyzed (Participants) | 327 | 318 | 645
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (15.3) | 57.2 (14.9) | 57.7 (16.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 187 | 355
  Male | 159 | 131 | 290
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 327 | 318 | 645

OUTCOME MEASURES:

1. Primary Outcome: Surgical Site Infection (SSI) Rate
Description: To evaluate the 30 day post-operative SSI rate in patients undergoing elective colorectal surgical procedures after intraoperative usage of Alexis O wound protector vs. CleanCision continuous irrigation wound protector.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Alexis O Wound Protector | CleanCision Wound Protector
Number analyzed (Participants) | 327 | 318
Participants
  Post-op Superficial SSI | 16 | 14
  Post-op Deep SSI | 6 | 1
  Post-op Organ/Space SSI | 6 | 3
  Composite Infection (SSIs + Wound Disruption) | 28 | 18

ADVERSE EVENTS:
Time Frame: 30 days following surgery
Arm/Group | Alexis O Wound Protector | CleanCision Wound Protector
All-Cause Mortality (participants affected / at risk) | 1/327 | 0/318
Serious Adverse Events (participants affected / at risk) | 0/327 | 0/318
Other Adverse Events (participants affected / at risk) | 98/327 | 95/318
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alexis O Wound Protector (N=327) | CleanCision Wound Protector (N=318)
Post-Op Sepsis (Infections and infestations) | 4 (4) | 2 (2)
Post-Op Pneumonia (Infections and infestations) | 2 (2) | 4 (4)
Post-Op Unplanned Intubation (General disorders) | 2 (2) | 0 (0)
Post-Op Deep Vein Thrombosis (Vascular disorders) | 3 (3) | 2 (2)
Post-Op Pulmonary Embolism (Vascular disorders) | 0 (0) | 1 (1)
Post-Op Acute Renal Failure (Renal and urinary disorders) | 1 (1) | 6 (6)
Post-Op Anastomotic Leak (Gastrointestinal disorders) | 1 (1) | 0 (0)
Post-Op C.Diff (Infections and infestations) | 4 (4) | 3 (3)
Post-Op Ileus (Gastrointestinal disorders) | 31 (31) | 26 (26)
Unplanned Reoperation (General disorders) | 7 (7) | 7 (7)
Readmission (Social circumstances) | 38 (38) | 36 (36)
Post-Op Urinary Tract Infection (Renal and urinary disorders) | 5 (5) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT03816995/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT03816995/ICF_001.pdf